CLINICAL TRIAL: NCT05612945
Title: Short-duration Aerobic High-intensity Intervals Versus Low-to-moderate-intensity Exercise Training in Symptomatic Patients With Peripheral Artery Disease: A Randomized Controlled Trial
Brief Title: High-intensity Intervals Versus Low-to-moderate-intensity Exercise Training in Patients With PAD
Acronym: HIIT_PAD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, Lucia Mazzolai, Prof, MD, PhD, Centre Hospitalier Universitaire Vaudois
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Exercise_intensity_PAD
Record Dates: First submitted 2022-10-31; First posted 2022-11-10 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Peripheral Arterial Disease
Keywords: Exercise; Rehabilitation; Physical activity
MeSH Terms: conditions — Peripheral Arterial Disease; Motor Activity

STUDY DESIGN:
Intervention Model Description: Monocentric randomized controlled trial (2 groups):
  Group 1 (n=30): high-intensity interval training group (HIIT) Group 2 (n=30): low-to-moderate intensity training group (LowMod)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-intensity interval training group (HIIT) (Experimental): Exercise training sessions will consist in an alternation of brief periods (≤ 60 s) of work performed at high intensity and brief period of passive rest.
  Patient will be asked to complete 1 set of 10-15x60-s (or 2 sets of 5-7x60-s) walking intervals. This protocol will elicits moderate-to-severe claudication pain during exertion. The training intensity in the HIIT group will be set at ≥85% HRpeak recorded during the maximal cardiopulmonary exercise test.
  Interventions: Other: High-intensity interval training group (HIIT)
- Low-to-moderate intensity training group (LowMod group) (Experimental): Exercise training sessions will consist in an alternation of periods of work performed at moderate exercise intensity and period of passive rest. The training approach of the LowMod group will be similar to the training prescription usually adopted in patients with claudication. The exercise training intensity will be set at ≤76% HRpeak recorded during the maximal cardiopulmonary exercise test.
  Interventions: Other: Low-to-moderate intensity training group (LowMod group)

INTERVENTIONS:
Other: High-intensity interval training group (HIIT) — Exercise training sessions will consist in an alternation of brief periods (≤ 60 s) of work performed at high intensity and brief period of passive rest.
  Patient will be asked to complete 1 set of 10-15x60-s (or 2 sets of 5-7x60-s) walking intervals. The training intensity in the HIIT group will be set at ≥85% HRpeak recorded during the maximal cardiopulmonary exercise test.
  The training intervention will consist of 36 walking sessions spread over 12 weeks. Each training session will lasted 30-60 min. The training intervention will be performed on a treadmill (Cosmed T150, Itlay), which is equipped with harness and chest belt to secure the patients and prevents falling. Each session started with a 5-min walking warm-up and ended with a 5min cool-down. During all the exercise training sessions, HR of the subjects will be continuously monitored (Polar M430, Finland).
  Arms: High-intensity interval training group (HIIT)
Other: Low-to-moderate intensity training group (LowMod group) — Exercise training sessions will consist in an alternation of periods of work performed at moderate exercise intensity and period of passive rest. The training approach of the LowMod group will be similar to the training prescription usually adopted in patients with claudication. The exercise training intensity will be set at ≤76% HRpeak recorded during the maximal cardiopulmonary exercise test.
  The training intervention will consist of 36 walking sessions spread over 12 weeks. Each training session will lasted 30-60 min. The training intervention will be performed on a treadmill (Cosmed T150, Itlay), which is equipped with harness and chest belt to secure the patients and prevents falling. Each session started with a 5-min walking warm-up and ended with a 5min cool-down. During all the exercise training sessions, HR of the subjects will be continuously monitored (Polar M430, Finland).
  Arms: Low-to-moderate intensity training group (LowMod group)

SUMMARY:
Supervised exercise training (SET) is considered among first-line therapies for patients with symptomatic lower extremity peripheral artery disease (PAD), combined with general cardiovascular risk management, lifestyle adaptation and pharmacological treatment.

Although without clear consistency, the guidelines give recommendations in terms of claudication pain severity, SET volume, duration, and frequency. However, no or little guidance is offered as far as training intensity is concerned. Most of the previous studies on SET, in the context of PAD, did not distinguish between symptom intensity and common training intensity measures such as % of maximal heart rate (%HRmax), % of HR reserve (%HRR), % of peak oxygen uptake (%VO2peak), % of VO2 reserve (%VO2R), or the rate of perceived exertion (RPE).

In a recent meta-analysis, we demonstrated that both training modality and exercise intensity (based on %peak heart rate, %peak oxygen uptake, or the rate of perceived exertion) should be considered when looking for the best results in patients with symptomatic PAD. These results call for study of the individual roles of each exercise intensity and modality on walking performance and cardiorespiratory fitness in patients with symptomatic PAD.

High-intensity interval training (HIIT) is composed of brief bursts of vigorous intensity interspersed with periods of rest or low-intensity exercise. HIIT may be better than moderate-intensity training (MIT) in improving cardiorespiratory fitness and functional capacity in patients with cardiovascular and metabolic diseases, but in patients with symptomatic PAD, the effects of such modalities on walking ability and cardiorespiratory fitness remain to be clearly determined.

The primary objective of this study is to compare the effects of 12-week-long exercise training (short-duration high-intensity intervals vs. low-to-moderate intensity) on treadmill performance in patients with symptomatic PAD.

It is hypothesized that treadmill performance would be improved to a greater extent after high-intensity exercise training

DETAILED DESCRIPTION:
Lower extremity peripheral artery disease (PAD) affects more than 200 million people worldwide. PAD is characterized by atherosclerotic lumen narrowing or occlusion of the lower limb arteries, leading to an imbalance between oxygen supply and demand downstream, especially in activated muscle during exertion. The hallmark symptom of PAD is typical intermittent claudication, defined as reproducible exertion-induced cramping or pain in the lower extremities, which is rapidly relieved with rest.

Patients with symptomatic PAD avoid exertion and tend to have muscle weakness, an altered gait and lower limb biomechanics. This results in impaired walking performance, accelerated functional decline, and reduced quality of life.

Supervised exercise training (SET) is considered among first-line therapies for patients with symptomatic PAD, combined with general cardiovascular risk management, lifestyle adaptation and pharmacological treatment. The clinical benefits of SET for patients with PAD are well established, with improved walking capacity and an improved quality of life as the primary outcomes.

Although without clear consistency, the guidelines give recommendations in terms of claudication pain severity, SET volume, duration, and frequency. However, no or little guidance is offered as far as training intensity is concerned. Most of the previous studies on SET, in the context of PAD, did not distinguish between symptom intensity and common training intensity measures such as % of maximal heart rate (%HRmax), % of HR reserve (%HRR), % of peak oxygen uptake (%VO2peak), % of VO2 reserve (%VO2R), or the rate of perceived exertion (RPE).

A meta-analysis by Parmenter et al. showed that vigorous (%HRpeak: 77-96, %VO2peak: 64-90, RPE: 14-17) exercise training improved cardiorespiratory fitness (VO2peak) more than light- to-moderate exercise therapy intensity in patients with PAD, but the changes in walking performance in these patients remain to be determined. In a recent meta-analysis, we demonstrated that both training modality and exercise intensity (based on %peak heart rate, %peak oxygen uptake, or the rate of perceived exertion) should be considered when looking for the best results in patients with symptomatic PAD. More precisely, we showed that, when training modalities were considered, walking at vigorous intensity showed the greatest improvement in maximal walking distance (MWD), while walking at light-to-moderate intensity showed the greatest improvement in pain-free walking distance. We also showed that vigorous was superior to light-to-moderate exercise intensity in improving cardiorespiratory fitness; and that, when training modalities were considered, cycling and other non-walking forms of training performed at vigorous intensity elicited the greatest improvements in cardiorespiratory fitness.

The results of our meta-analysis call for study of the individual roles of each exercise intensity and modality on walking performance and cardiorespiratory fitness in patients with symptomatic PAD.

High-intensity interval training (HIIT) is composed of brief bursts of vigorous intensity interspersed with periods of rest or low-intensity exercise. HIIT may be better than moderate-intensity training (MIT) in improving cardiorespiratory fitness and functional capacity in patients with cardiovascular and metabolic diseases, but in patients with symptomatic PAD, the effects of such modalities on walking ability and cardiorespiratory fitness remain to be clearly determined.

The primary objective of this study is to compare the effects of 12-week-long exercise training (short-duration high-intensity intervals vs. low-to-moderate intensity) on treadmill performance in patients with symptomatic PAD.

It is hypothesized that treadmill performance would be improved to a greater extent after high-intensity exercise training

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with symptomatic PAD (Fontaine stage IIa/b);
* ABI ≤ 0.9 or drop by 20% following exercise treadmill test 1;
* TBI ≤ 0.6 if incompressible arteries (diabetes and renal insufficiency);
* Signed written informed consent form.

Exclusion Criteria:

* Age < 18;
* Unable to walk at 3.2 km/h on a treadmill (slope 0%) at least 300 m;
* Previous participate in SET programs ≤ 1 year;
* Prior leg/foot amputation;
* Contraindication to exercise
* Neurological and neuromuscular disorders and other comorbidities (orthopedic, rheumatologic) leading to gait abnormalities.
* Known Pregnancy
* Incapacity of discernment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Maximal walking distance | This will be assessed before and after the 3-month training program. The post-program assessment will be performed between 5 to 14 days following the last training session.
  Patients will perform an incremental treadmill test to determine the maximal walking distance (MWD). Initial walking speed will be set at 3.2 km/h, and at 0% grade. The grade will be increased by 2% each 2 min.

SECONDARY OUTCOMES:
Functional performance - 6-minute walk test | This will be assessed before and after the 3-month training program. The post-program assessment will be performed between 5 to 14 days following the last training session.
  Patients will perform the 6-minute walk test
Functional performance - ascending and descending stair performance test | This will be assessed before and after the 3-month training program. The post-program assessment will be performed between 5 to 14 days following the last training session.
  Patients will perform the ascending and descending stair performance test
Functional performance - short physical performance battery test | This will be assessed before and after the 3-month training program. The post-program assessment will be performed between 5 to 14 days following the last training session.
  Patients will perform the short physical performance battery test
Functional performance - preferred walking speed and gait analysis assessment | This will be assessed before and after the 3-month training program. The post-program assessment will be performed between 5 to 14 days following the last training session.
  Patients will perform the preferred walking speed and gait analysis assessment
Functional performance - unipedal stance test | This will be assessed before and after the 3-month training program. The post-program assessment will be performed between 5 to 14 days following the last training session.
  Patients will perform the unipedal stance test
Functional performance - 30- and 60-s repeated sit-to-stand chair test | This will be assessed before and after the 3-month training program. The post-program assessment will be performed between 5 to 14 days following the last training session.
  Patients will perform the 30- and 60-s repeated sit-to-stand chair test.
Cardiorespiratory fitness (VO2peak) | This will be assessed before and after the 3-month training program. The post-program assessment will be performed between 5 to 14 days following the last training session.
  Patients will perform a maximal cardiopulmonary exercise test
Muscle oxygenation during treadmill test | This will be assessed before and after the 3-month training program. The post-program assessment will be performed between 5 to 14 days following the last training session.
  Muscle oxygenation will be assessed during treadmill test by near-infrared spectroscopy (NIRS)
Hemodynamic parameters | This will be assessed before and after the 3-month training program. The post-program assessment will be performed between 5 to 14 days following the last training session.
  Ankle - toe brachial index (ABI, TBI)
Self-perceived quality of life and walking (dis)abilities | This will be assessed before and after the 3-month training program. The post-program assessment will be performed between 5 to 14 days following the last training session.
  Self-perceived quality of life (Medical Outcomes Study Short-Form 36 (SF-36) and walking (dis)abilities (Walking Impairement Questionnaire, WIQ) will be assessed. Each questionnaire has scores on a 0-100 scale (0 (worse score) to 100 (best score)).
Total amount of physical activity | This will be assessed before and after the 3-month training program. The post-program assessment will be performed between 5 to 14 days following the last training session.
  The total amount of physical activity will be assessed by accelerometer.
Pain-free walking distance | This will be assessed before and after the 3-month training program. The post-program assessment will be performed between 5 to 14 days following the last training session.
  Patients will perform an incremental treadmill test to determine the pain-free walking distance (PFWD). Initial walking speed will be set at 3.2 km/h, and at 0% grade. The grade will be increased by 2% each 2 min.

CONTACTS AND LOCATIONS:
Locations (1):
- CHUV, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.

REFERENCES:
- [Derived] Lanzi S, Pousaz A, Fresa M, Besson C, Desgraz B, Gremeaux-Bader V, Mazzolai L. Short-duration aerobic high-intensity intervals versus moderate exercise training intensity in patients with peripheral artery disease: study protocol for a randomised controlled trial (the Angiof-HIIT Study). BMJ Open. 2024 Apr 17;14(4):e081883. doi: 10.1136/bmjopen-2023-081883. PMID 38631833